CLINICAL TRIAL: NCT07290556
Title: Establishing the Preliminary Utility of a Novel Pediatric Manual Mobile Standing Wheelchair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Optimal Mobility, Inc (Industry)
Collaborators: Gillette Children's Specialty Healthcare (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00086649; R44HD118822 (NIH)
Record Dates: First submitted 2025-11-25; First posted 2025-12-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Spina Bifida
Keywords: Spinal Bifida; Wheelchair; Pediatric; Standing
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experiment 1: In-Lab Testing (Experimental): Perform tasks in a laboratory environment designed to test the maneuverability and ease of use of the PedMMSWC as compared to commercial devices.
  Interventions: Device: PedMMSWC Wheelchair User Testing
- Experiment 2: Simulated Community and Home Testing (Experimental): Perform tasks in a simulated home, school, and community setting using the PedMedWC wheelchair.
  Interventions: Device: PedMMSWC Simulated Home, School, Community Environment

INTERVENTIONS:
Device: PedMMSWC Wheelchair User Testing — The PedMMSWC standing wheelchair prototype will be tested and compared with a standing frame during Experiment 1: In-Lab Testing.
  Arms: Experiment 1: In-Lab Testing
Device: PedMMSWC Simulated Home, School, Community Environment — The PedMMSWC standing wheelchair will be tested in a simulated home, school, and community environment. Participants will be given assigned tasks and be scored on completion of activities.
  Arms: Experiment 2: Simulated Community and Home Testing

SUMMARY:
To establish the preliminary utility of a novel pediatric manual mobile standing wheelchair (PedMMSWC).

ELIGIBILITY:
Inclusion Criteria:

* 8 - 17 years old
* Primarily use a manual wheelchair for daily mobility
* Are actively enrolled in a standing program
* Fit the height and weight requirements of the PedMMSWC
* Can follow simple verbal instructions
* Are able to speak and read in English

Exclusion Criteria:

* Have insufficient trunk control to maneuver in seated and standing positions
* Have lower limb contracture which would preclude standing
* Have had orthopedic surgery within the last twelve months
* Have pressure injuries at the location where the PedMMSWC interfaces
* Have insufficient fine motor skills to independently initiate the sit-to-stand function
* Have a history of uncontrolled seizures or cardiovascular conditions that would make participation unsafe

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-08-25 (Estimated); Study Completion 2027-08-25 (Estimated)

PRIMARY OUTCOMES:
Comparison of a modified Wheelchair Skills Test with Participants wheelchair to the PedMMSWC | Day 1
  The primary outcome measure for this aim is user performance on a modified Wheelchair Skills Test (mWST) under three test conditions: PedMMSWC in the seated position, PedMMSWC in the standing position, and the individuals' daily wheelchair.
  The investigators hypothesize that performance on the mWST in the PedMMSWC will not be clinically inferior to performance in individuals' daily wheelchairs.

SECONDARY OUTCOMES:
100-Meter Roll Test (meters per second) | Day 1
  Participants will perform a 100-meter roll test in the PedMMSWC (in seated and standing) and their daily wheelchair (dWC). This test is originally described in the WST Version 4.1 and measures how quickly (meters per second) participants can cover 100 meters in their wheelchair over hard, flat, level ground. Participants will perform the test once in each device condition (PedMMSWC-Seated, PedMMSWC-Standing, dWC), rate their perceived exertion, and speed following each test.
100-Meter Roll Test (perceived exertion) | Day 1
  Participants will perform a 100-meter roll test in the PedMMSWC (in seated and standing) and their daily wheelchair (dWC). This test measures how much effort (percieved exertion) participants use to cover 100 meters in their wheelchair over hard, flat, level ground. Participants will perform the test once in each device condition (PedMMSWC-Seated, PedMMSWC-Standing, dWC) and rate their perceived exertion.
Pressure Mapping (peak pressure (mm/hg)) | Day 1
  Participants will be measured with a pressure mapping device for peak pressure (mm/hg) in the PedMMSWC sitting, PedMMSWC standing, and the Easy Stand Device on interfacing surfaces.
Pressure Mapping (coefficient of variation) | Day 1
  Participants will be measured with a pressure mapping device for coefficient of variation in the PedMMSWC sitting, PedMMSWC standing, and the Easy Stand Device on interfacing surfaces.
Functional Mobility Assessment - Family Centered (FMA-FC) | Day 1 or 2
  To capture baseline satisfaction with individuals' primary wheelchair, each participant and their caregiver will collaboratively complete the FMA-FC outcome measure, which has been specifically designed and validated for pediatric use.
Participant and Caregiver Perceptions of Device | Day 1 or Day 2
  Participants will complete a course in the PedMMSWC and their dWC designed to simulate typical activities in home, school, and community environments. In each of these environments, participants will engage in a series of structured activities tailored to their developmental level. While using the PedMMSWC, participants will also complete a 'free play' period during which they will be encouraged to explore and spontaneously interact with the space. Individuals will have free choice to move between seated and standing positions in the PedMMSWC for all tasks and play. Outcomes: qualitative and coded interview data, why and how often sit-to-stand transitions occur, the time spent standing, and therapist score task completion and safety on a 4-point scale.

OTHER OUTCOMES:
User-Device Movement during Sit-to-Stand Transitions (degrees of motion) | Day 1
  Using body motion analysis, investigators will record and analyze sit-to-stand transitions in a standing frame and the PedMMSWC wheelchair. Measuring three dimensional rotation of the thigh, shank, torso segments relative to the wheelchair during sit to stand transitions. during sit-to-stand transitions.
User-Device Movement during Sit-to-Stand Transitions (mm) | Day 1
  Using body motion analysis, investigators will record and analyze sit-to-stand transitions in a standing frame and the PedMMSWC wheelchair. Measuring the offset and translation (mm) of the body segments (trunk and thigh) relative to the chair or standing frame during sit-to-stand transitions.
User-Device Movement during Sit-to-Stand Transitions (seconds) | Day 1
  Using body motion analysis, investigators will record and analyze sit-to-stand transitions in a standing frame and the PedMMSWC wheelchair. Measuring time-to-stand (seconds), time-to-sit (seconds) in the chair or standing frame during sit-to-stand transitions.

CONTACTS AND LOCATIONS:
Locations (1):
- Gillette Children's Specialty Healthcare, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Company (sponsor) Website — https://optimal-mobility.com/